CLINICAL TRIAL: NCT00558428
Title: An Eight-week Randomized, 4-arm, Double-blind Study to Compare the Efficacy and Safety of Combinations of Telmisartan 40mg + Amlodipine 5mg Versus Telmisartan 80mg + Amlodipine 5mg Versus Amlodipine 5mg Versus Amlodipine 10mg Monotherapy in Patients With Hypertension Who Fail to Respond Adequately to Treatment With Amlodipine 5mg Monotherapy
Brief Title: Telmisartan/Amlodipine (80/5) vs. Telmisartan/Amlodipine (40/5) vs. Amlodipine 10 or 5 in Resistant Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1235.5; EUDRACT2007-002409-36
Record Dates: First submitted 2007-10-29; First posted 2007-11-15 (Estimated); Results first posted 2009-12-15 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

INTERVENTIONS:
Drug: fixed dose combination of telmisartan+amlodipine
Drug: amlodipine

SUMMARY:
The primary objectives of this trial are (a) to demonstrate that the fixed-dose combination T40/A5 or the fixed-dose combination T80/A5 is superior in reducing blood pressure at eight weeks compared with A5 (b) to demonstrate that the fixed-dose combination T40/A5 or the fixed-dose combination T80/A5 is not inferior in reducing blood pressure at eight weeks compared with A10 and (c) to demonstrate that the incidence of oedema on the fixed-dose combination T40/A5 pooled with the fixed-dose combination T80/A5 is superior (less oedema) to A10 in patients who fail to respond adequately to six weeks treatment with A5.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged at least 18 years at the date of signing the consent form
2. diagnosis of essential hypertension and blood pressure not adequately controlled before enrolment in the study
3. failure to respond adequately to six weeks treatment with amlodipine 5 mg monotherapy
4. able to stop any current antihypertensive therapy without unacceptable risk to the patient (Investigator's decision)
5. willing and able to provide written informed consent (in accordance with Good Clinical Practice and local legislation).

Exclusion Criteria:

1. are not practising acceptable means of birth control or do not plan to continue using acceptable means of birth control throughout the study and do not agree to submit to pregnancy testing during participation in the trial. Acceptable methods of birth control include the transdermal patch, oral, implantable or injectable contraceptives, sexual abstinence and vasectomised partner.
2. known or suspected secondary hypertension
3. mean seated systolic blood pressure (SBP) over 200 mmHg and/or mean seated diastolic blood pressure (DBP) over 120 mmHg at Visit 1 or 2 or mean seated SBP over 180 mmHg and/or mean seated DBP over 120 mmHg at the end of the run-in period (Visit 3)
4. any clinically significant hepatic impairment (e.g. clinically significant cholestasis, biliary obstructive disorder or hepatic insufficiency)
5. severe renal impairment (e.g. serum creatinine >3.0 mg/dL or >265 mcmol/L, known creatinine clearance <30mL/min or clinical markers of severe renal impairment)
6. bilateral renal artery stenosis or renal artery stenosis in a solitary kidney or post-renal transplant
7. clinically relevant hyperkalaemia
8. uncorrected volume or sodium depletion.
9. primary aldosteronism.
10. hereditary fructose or lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1098 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (129):
- Belgium (9):
  - 1235.5.32004 Boehringer Ingelheim Investigational Site, Aywaille
  - 1235.5.32001 Boehringer Ingelheim Investigational Site, Brussels
  - 1235.5.32010 Boehringer Ingelheim Investigational Site, Gozée
  - 1235.5.32008 Boehringer Ingelheim Investigational Site, Linkebeek
  - 1235.5.32003 Boehringer Ingelheim Investigational Site, Mol
  - 1235.5.32007 Boehringer Ingelheim Investigational Site, Natoye
  - 1235.5.32009 Boehringer Ingelheim Investigational Site, Tavier
  - 1235.5.32002 Boehringer Ingelheim Investigational Site, Tienen-Kumtich
  - 1235.5.32005 Boehringer Ingelheim Investigational Site, Turnhout
- Canada (12):
  - 1235.5.20001 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1235.5.20011 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1235.5.20007 Boehringer Ingelheim Investigational Site, Bay Roberts, Newfoundland and Labrador
  - 1235.5.20005 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 1235.5.20008 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1235.5.20013 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1235.5.20014 Boehringer Ingelheim Investigational Site, Etobicoke, Ontario
  - 1235.5.20010 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1235.5.20012 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1235.5.20009 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1235.5.20006 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1235.5.20003 Boehringer Ingelheim Investigational Site, Sainte-Foy, Quebec
- Denmark (8):
  - 1235.5.45002 Boehringer Ingelheim Investigational Site, Birkerød
  - 1235.5.45005 Boehringer Ingelheim Investigational Site, Haderslev
  - 1235.5.45008 Boehringer Ingelheim Investigational Site, Herning
  - 1235.5.45009 Boehringer Ingelheim Investigational Site, Hinnerup
  - 1235.5.45001 Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - 1235.5.45006 Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - 1235.5.45003 Boehringer Ingelheim Investigational Site, Vaerløse
  - 1235.5.45007 Boehringer Ingelheim Investigational Site, Vildbjerg
- Finland (4):
  - 1235.5.35003 Boehringer Ingelheim Investigational Site, Joensuu
  - 1235.5.35004 Boehringer Ingelheim Investigational Site, Joensuu
  - 1235.5.35001 Boehringer Ingelheim Investigational Site, Turku
  - 1235.5.35002 Boehringer Ingelheim Investigational Site, Turku
- France (50):
  - 1235.5.3301H Boehringer Ingelheim Investigational Site, Aigrefeuille S/Maine
  - 1235.5.3306C Boehringer Ingelheim Investigational Site, Angers
  - 1235.5.3309B Boehringer Ingelheim Investigational Site, Angers
  - 1235.5.3309C Boehringer Ingelheim Investigational Site, Angers
  - 1235.5.3309E Boehringer Ingelheim Investigational Site, Angers
  - 1235.5.3309D Boehringer Ingelheim Investigational Site, Avrillé
  - 1235.5.3309A Boehringer Ingelheim Investigational Site, Beaucouzé
  - 1235.5.3303B Boehringer Ingelheim Investigational Site, Bono
  - 1235.5.3305A Boehringer Ingelheim Investigational Site, Bourg Des Cptes
  - 1235.5.3306D Boehringer Ingelheim Investigational Site, Briollay
  - 1235.5.3308B Boehringer Ingelheim Investigational Site, Cholet
  - 1235.5.3308C Boehringer Ingelheim Investigational Site, Cholet
  - 1235.5.3308D Boehringer Ingelheim Investigational Site, Cholet
  - 1235.5.3308F Boehringer Ingelheim Investigational Site, Cholet
  - 1235.5.3302C Boehringer Ingelheim Investigational Site, Garchizy
  - 1235.5.3303C Boehringer Ingelheim Investigational Site, Grandchamps
  - 1235.5.3302D Boehringer Ingelheim Investigational Site, Guérigny
  - 1235.5.3310A Boehringer Ingelheim Investigational Site, Jarny
  - 1235.5.3301L Boehringer Ingelheim Investigational Site, La Chapelle /s Erdre
  - 1235.5.3301J Boehringer Ingelheim Investigational Site, La Chapelle-sur-Erdre
  - 1235.5.3304A Boehringer Ingelheim Investigational Site, La Fresnais
  - 1235.5.3308E Boehringer Ingelheim Investigational Site, La Jubaudière
  - 1235.5.3301G Boehringer Ingelheim Investigational Site, La Montagne
  - 1235.5.3307D Boehringer Ingelheim Investigational Site, Le Mesnil-en-Vallée
  - 1235.5.3301E Boehringer Ingelheim Investigational Site, Le Temple-de-Bretagne
  - 1235.5.3309F Boehringer Ingelheim Investigational Site, Les Ponts-de-Cé
  - 1235.5.3307G Boehringer Ingelheim Investigational Site, Loudun
  - 1235.5.3305B Boehringer Ingelheim Investigational Site, Louvigné Le Bais
  - 1235.5.3307E Boehringer Ingelheim Investigational Site, Mouliherne
  - 1235.5.3306A Boehringer Ingelheim Investigational Site, Mûrs-Erigné
  - 1235.5.3307A Boehringer Ingelheim Investigational Site, Mûrs-Erigné
  - 1235.5.3301A Boehringer Ingelheim Investigational Site, Nantes
  - 1235.5.3301B Boehringer Ingelheim Investigational Site, Nantes
  - 1235.5.3301D Boehringer Ingelheim Investigational Site, Nantes
  - 1235.5.3301M Boehringer Ingelheim Investigational Site, Nantes
  - 1235.5.3302A Boehringer Ingelheim Investigational Site, Nevers
  - 1235.5.3302F Boehringer Ingelheim Investigational Site, Nevers
  - 1235.5.3301I Boehringer Ingelheim Investigational Site, Nort-sur-Erdre
  - 1235.5.3301C Boehringer Ingelheim Investigational Site, Orvault
  - 1235.5.3307F Boehringer Ingelheim Investigational Site, Parçay-les-Pins
  - 1235.5.3301F Boehringer Ingelheim Investigational Site, Saint Aubin Les Châteaux
  - 1235.5.3306F Boehringer Ingelheim Investigational Site, Saint-Georges-de-Montaigu
  - 1235.5.3304B Boehringer Ingelheim Investigational Site, Saint-Ouen-la-Rouërie
  - 1235.5.3307C Boehringer Ingelheim Investigational Site, Saint-Pierre-Montlimart
  - 1235.5.3301N Boehringer Ingelheim Investigational Site, Sautron
  - 1235.5.3306B Boehringer Ingelheim Investigational Site, Segré
  - 1235.5.3306E Boehringer Ingelheim Investigational Site, Thouars
  - 1235.5.3304C Boehringer Ingelheim Investigational Site, Tinténiac
  - 1235.5.3303A Boehringer Ingelheim Investigational Site, Vannes
  - 1235.5.3308A Boehringer Ingelheim Investigational Site, Vihiers
- Netherlands (8):
  - 1235.5.31008 Boehringer Ingelheim Investigational Site, Beerzerveld
  - 1235.5.31006 Boehringer Ingelheim Investigational Site, Bennebroek
  - 1235.5.31004 Boehringer Ingelheim Investigational Site, Hoogwoud
  - 1235.5.31003 Boehringer Ingelheim Investigational Site, Musselkanaal
  - 1235.5.31007 Boehringer Ingelheim Investigational Site, Nijverdal
  - 1235.5.31001 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1235.5.31005 Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - 1235.5.31010 Boehringer Ingelheim Investigational Site, Voerendaal
- Norway (4):
  - 1235.5.47001 Boehringer Ingelheim Investigational Site, Ålesund
  - 1235.5.47002 Boehringer Ingelheim Investigational Site, Bergen
  - 1235.5.47003 Boehringer Ingelheim Investigational Site, Hamar
  - 1235.5.47004 Boehringer Ingelheim Investigational Site, Oslo
- Philippines (8):
  - 1235.5.63006 Boehringer Ingelheim Investigational Site, Makati City
  - 1235.5.63001 Boehringer Ingelheim Investigational Site, Manila
  - 1235.5.63002 Boehringer Ingelheim Investigational Site, Manila
  - 1235.5.63009 Boehringer Ingelheim Investigational Site, Manila
  - 1235.5.63008 Boehringer Ingelheim Investigational Site, Pasay
  - 1235.5.63005 Boehringer Ingelheim Investigational Site, Pasig
  - 1235.5.63003 Boehringer Ingelheim Investigational Site, Quezon City
  - 1235.5.63007 Boehringer Ingelheim Investigational Site, Quezon City
- South Africa (9):
  - 1235.5.27003 Boehringer Ingelheim Investigational Site, Boksburg
  - 1235.5.27006 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.5.27009 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.5.27010 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.5.27004 Boehringer Ingelheim Investigational Site, Durban
  - 1235.5.27008 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1235.5.27001 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 1235.5.27005 Boehringer Ingelheim Investigational Site, Lenasia
  - 1235.5.27002 Boehringer Ingelheim Investigational Site, Pretoria
- South Korea (8):
  - 1235.5.82007 Boehringer Ingelheim Investigational Site, Busan
  - 1235.5.82001 Boehringer Ingelheim Investigational Site, Daegu
  - 1235.5.82006 Boehringer Ingelheim Investigational Site, Daejeon
  - 1235.5.82004 Boehringer Ingelheim Investigational Site, Gangwon-Do
  - 1235.5.82008 Boehringer Ingelheim Investigational Site, Gwangju
  - 1235.5.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.5.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.5.82005 Boehringer Ingelheim Investigational Site, Seoul
- Sweden (5):
  - 1235.5.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1235.5.46003 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1235.5.46005 Boehringer Ingelheim Investigational Site, Luleå
  - 1235.5.46004 Boehringer Ingelheim Investigational Site, Rättvik
  - 1235.5.46001 Boehringer Ingelheim Investigational Site, Stockholm
- Taiwan (4):
  - 1235.5.88605 Boehringer Ingelheim Investigational Site, Changhua
  - 1235.5.88608 Boehringer Ingelheim Investigational Site, Hualien City
  - 1235.5.88601 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1235.5.88603 Boehringer Ingelheim Investigational Site, Taichung

REFERENCES:
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/1235/1235.5_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1487 were enrolled, 1098 entered but 1 patient not treated.
Period: Overall Study
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Started | 267 | 276 | 277 | 277
Completed | 255 | 252 | 273 | 266
Not Completed | 12 | 24 | 4 | 11
Not completed — Adverse Event | 6 | 22 | 3 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2
Not completed — Non compliant with protocol | 1 | 0 | 0 | 3
Not completed — Consent withdrawn | 2 | 1 | 0 | 1
Not completed — Other | 3 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Total
Number analyzed (Participants) | 267 | 276 | 277 | 277 | 1097
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (10.6) | 54.3 (10.6) | 53.9 (11) | 54.5 (10.2) | 54.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 100 | 117 | 94 | 415
  Male | 163 | 176 | 160 | 183 | 682

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Seated Diastolic Blood Pressure (DBP)
Description: Change from baseline to the end of study in trough DBP
Time Frame: End of study (8 weeks or last value on treatment)
Population: Full analysis set of patients who had a baseline trough blood pressure measurement and at least one post baseline trough blood pressure measurement using last observation carried forward. The full analysis set included patients who had baseline and at least one post baseline trough measure of blood pressure
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Number analyzed (Participants) | 255 | 261 | 270 | 271
mmHg | -5.71 (0.49) | -7.95 (0.49) | -9.35 (0.48) | -10.63 (0.48)
Statistical Analysis 1: Comparison: Amlodipine 5mg vs Telmisartan 40mg and Amlodipine 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted for baseline and country effect; Least Squares Mean Difference = -3.64, 95% CI [-4.90 to -2.38], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Amlodipine 5mg vs Telmisartan 80mg and Amlodipine 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted for baseline and country effect; Least Squares Mean Difference = -4.92, 95% CI [-6.18 to -3.66], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Amlodipine 10mg vs Telmisartan 40mg and Amlodipine 5mg; Test type: Superiority or Other; ANCOVA; Adjusted for baseline and country effect; Least Squares Mean Difference = -1.40, 95% CI [-2.66 to -0.14], Standard Error of Mean 0.64
Statistical Analysis 4: Comparison: Amlodipine 10mg vs Telmisartan 80mg and Amlodipine 5mg; Test type: Superiority or Other; ANCOVA; Adjusted for baseline and country effect; Least Squares Mean Difference = -2.68, 95% CI [-3.93 to -1.43], Standard Error of Mean 0.64

2. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure (SBP)
Description: Change from baseline to the end of study in trough SBP
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Number analyzed (Participants) | 255 | 261 | 270 | 271
mmHg | -6.18 (0.73) | -11.11 (0.72) | -13.56 (0.71) | -14.99 (0.71)

3. Secondary Outcome: Trough Seated Diastolic Blood Pressure Control
Description: The number of patients who reach the target DBP of <90mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Number analyzed (Participants) | 255 | 261 | 270 | 271
patients
  Yes (DBP<90 mmHg) | 107 | 148 | 153 | 173
  No (DBP>=90 mmHg) | 148 | 113 | 117 | 98

4. Secondary Outcome: Trough Seated DBP Response
Description: The number of patients who reach the target DBP of <90mmHg or had a reduction in DBP >= 10mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Number analyzed (Participants) | 255 | 261 | 270 | 271
patients
  Yes (Responder) | 116 | 163 | 177 | 187
  No (Non-responder) | 139 | 98 | 93 | 84

5. Secondary Outcome: Trough Seated SBP Control
Description: The number of patients who reach the target SBP of <140mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Number analyzed (Participants) | 255 | 261 | 270 | 271
patients
  Yes (SBP<140 mmHg) | 100 | 142 | 162 | 178
  No (SBP>=140 mmHg) | 155 | 119 | 108 | 93

6. Secondary Outcome: Trough Seated SBP Response
Description: The number of patients who reach the target SBP of <140mmHg or had a reduction in SBP >= 15 mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Number analyzed (Participants) | 255 | 261 | 270 | 271
patients
  Yes (Responder) | 118 | 166 | 187 | 200
  No (Non-responder) | 137 | 95 | 83 | 71

7. Secondary Outcome: Trough Seated Blood Pressure (BP) Normality Classes
Description: The number of patients who reach predefined BP categories:
  * Optimal - SBP<120 and DBP<80 mmHg
  * Normal - SBP<130 and DBP<85 mmHg
  * High-normal - SBP<140 DBP<90 mmHg
  * Stage 1 hypertension - SBP<160 and DBP<100
  * Stage 2 hypertension SBP>=160 and DBP>=100 mmHg
Time Frame: End of study (8 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: patients
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Number analyzed (Participants) | 255 | 261 | 270 | 271
patients
  Optimal | 2 | 5 | 19 | 21
  Normal | 23 | 30 | 35 | 51
  High-normal | 42 | 68 | 63 | 67
  Stage 1 hypertension | 118 | 126 | 127 | 110
  Stage 2 hypertension | 70 | 32 | 26 | 22

8. Primary Outcome: Number of Patients With Oedema
Description: Patients from the treated set who experienced at least one case of general oedema.
Time Frame: During randomised treatment period (8 weeks was the planned end of treatment, some of the measurements analysed as end of study can be at 4 weeks or at any point on randomised treatment)
Population: The treated set (TS) consisted of all patients that took at least one dose of the double-blind treatment (n=1097)
Measure: Number; unit: patients
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Number analyzed (Participants) | 255 | 261 | 270 | 271
patients
  Number of patients with any oedema | 23 | 76 | 14 | 10
  Number of patients with general oedema | 23 | 75 | 14 | 10

ADVERSE EVENTS:
Time Frame: From day of first dose until one day after last dose
Arm/Group | Amlodipine 5mg | Amlodipine 10mg | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Serious Adverse Events (participants affected / at risk) | 2/267 | 1/276 | 2/277 | 1/277
Other Adverse Events (participants affected / at risk) | 22/267 | 74/276 | 14/277 | 10/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine 5mg (N=267) | Amlodipine 10mg (N=276) | Telmisartan 40mg and Amlodipine 5mg (N=277) | Telmisartan 80mg and Amlodipine 5mg (N=277)
Atrial fibrilation (Cardiac disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine 5mg (N=267) | Amlodipine 10mg (N=276) | Telmisartan 40mg and Amlodipine 5mg (N=277) | Telmisartan 80mg and Amlodipine 5mg (N=277)
Oedema peripheral (General disorders) | 22 | 74 | 14 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.